CLINICAL TRIAL: NCT05012514
Title: Effects of Led Photobiomodulation Therapy on the Subcutaneous Fatty Tissue of Obese Individuals- Histological and Immunohistochemical Analysis
Brief Title: Effects of Led Photobiomodulation Therapy
Acronym: LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLLT
Record Dates: First submitted 2021-08-03; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Photobiomodulation

STUDY DESIGN:
Intervention Model Description: Participants received seven sessions of PBMT LED twice a week, the last session being about twenty minutes before the surgical procedure of bariatric surgery. The therapy was performed on the left side of the abdominal region following the linea alba of all research participants and the right side was considered as control, for application they will receive eye protection, using goggles for safety, the abdomen of the participants will be cleaned by using a neutral cleansing soap.
Masking Description: N/D
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control- Without intervention (No Intervention): The participants have the right side of the abdomen as a control without inversion
- LLLT- With intervention (Active Comparator): The participants received the LED PBMT treatment with associated red and infrared wavelengths sequentially on the left side of the abdomen
  Interventions: Device: LLLT RED

INTERVENTIONS:
Device: LLLT RED — Participants received seven sessions of PBMT LED twice a week, the last session being about twenty minutes before the surgical procedure of bariatric surgery. The therapy was performed on the left side of the abdominal region following the linea alba of all research participants and the right side was considered as control, for application they will receive eye protection, using goggles for safety, the abdomen of the participants will be cleaned by using a neutral cleansing soap. A cluster applicator was used using the parameters described in table 1.
  For therapy, the equipment Antares® was used, IBRAMED- Indústria Brasileira de Equipamentos Eletromédicos EIRELI [EIRELI Brazilian Industry of Electromedical Equipment], approved by Anvisa Nº 10360310037. Figure 1.
  Arms: LLLT- With intervention

SUMMARY:
Background: Photobiomodulation therapy (PBMT) has become an adjuvant therapeutic possibility in body remodeling procedures. Although this modality emerged in 1960, there are still few studies that demonstrate the real mechanism of action and possible interaction with subcutaneous fatty tissue. Given this scenario, this study was proposed with the aim of evaluating the effects of PBMT to Light Emitting Diode (LED) associating the red (630 nm) and infrared (850 nm) wavelengths in the subcutaneous fatty tissue. Methods: This is a non-randomized controlled study of comparative intervention that evaluated a sample of subcutaneous fatty tissue from women with grade II obesity. The participants received the LED PBMT treatment with associated red and infrared wavelengths sequentially on the left side of the abdomen and the right side was considered as control, with the collection of biological material performed at the time of bariatric surgery. For histological and immunohistochemical evaluation, Caspase 3, Cleaved Caspase 3, CD68+, HSL and adipophilin markers were used.

DETAILED DESCRIPTION:
Localized adiposity or localized obesity is the hyperplasia or hypertrophy of adipocytes in specific areas such as the abdomen and flanks, its development is associated with the risk of metabolic diseases and psychosocial changes related to low self-esteem, since aesthetic appearance is considered an imposed standard of beauty nowadays.

The proportion of obese individuals has increased at alarming levels around the world and to combat it, several therapeutic approaches are needed, such as personalized diets and physical activity plans, in order to balance consumption and energy expenditure, but despite these controls, several adjuvant features such as non-invasive modalities are also being proposed to reduce subcutaneous fatty tissue.

Among these modalities are the technologies of shock waves, cryolipolysis, focused ultrasound, radiofrequency and the use of light sources with photobiomodulation therapy. The latter, in turn, has shown relevant results in the possible reduction of subcutaneous fatty tissue.

The use of a light source as a therapeutic form is already millenary and nowadays it is widely used as a modality to promote wound healing, reduce pain and possible damage and inflammation of tissues with the characteristic of not presenting photothermal or photoacoustic effects, thus termed as photobiomodulation therapy (PBMT). It can be used by using non-ionizing light sources such as Low Intensity Laser Therapy (LLLT) or Light Emitting Diode Therapy (LED).

The landmark of the use of PBMT in the possible reduction of subcutaneous fatty tissue emerged with the double-blind randomized placebo-controlled study by Jackson et al. in 2012. A total of 689 individuals participated in the study, subdivided into a placebo group and an LLLT group, all of whom were evaluated during the treatment, in order to verify the possible reduction in the circumference of the waist, hips and thighs. Participants received a total of six LLLT treatments over 2 weeks with baseline and post-procedure circumferential measurements recorded. The results showed a significant reduction (p<0.0001) in circumference at the waist, hips and thighs one week after treatment with LLLT.

Following the same line of research Jankowski et al., and Elnaggar, also carried out photobiomodulation studies to reduce fatty tissue and show partially significant results. The justification for the result was the smaller sample of participants compared to the study by Jackson et al., , however these studies were not able to elucidate which form of therapeutic action on fatty tissue to promote its reduction.

The mechanisms by which PBMT can affect fatty tissue are still controversial, and it is hypothesized that PBMT could induce micropores in the adipocyte membrane, which allow the release of intracellular lipids and place them outside the interstitial space or an alternative hypothesis is that PBMT stimulates mitochondria in adipocytes, which, in turn, increases adenosine triphosphate (ATP) synthesis with subsequent activation of cyclic adenosine monophosphate (cAMP), promoting lipolysis, and the third hypothesis is that it depends on of the dose applied in PBMT, this can even stimulate adipocyte cell apoptosis, that is, there is still no clear physiological basis for its mechanism.

Another important PBMT fact for the reduction of fatty tissue observed in articles already published is the difference in the wavelengths used, and in some articles the photobiomodulation was carried out with the red wavelength 630nm and in others the infrared 808 or 850nm. It is believed that each of them must reach different depths of the fatty tissue and thus favor its reduction, however, there is no standardization of the protocol.

Given this scenario, this study aimed to verify the real mechanism of action of PBMT when used in association of the wavelengths, red (630nm) and infrared (850nm) in the subcutaneous fatty tissue, through a clinical study with histological and immunohistochemistry analysis with markers of lipolysis and apoptosis in the subcutaneous fatty tissue of obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* As inclusion criteria, women participating in the group of pre-surgical preparation for bariatric surgery at the Hospital de Clínicas da Unicamp [Unicamp Clinics Hospital], presenting obesity degrees II and III, who had weight loss of at least 10% of the initial weight with indication for bariatric surgery.

Exclusion Criteria:

* As exclusion criteria, women presenting diabetes mellitus, with skin lesions such as dermatitis and dermatosis, with a history of deep venous thrombosis, smokers, or who had electronic implanted devices such as cardiac pacemakers were ineligible.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
immunohistochemical evaluation | one month
  immunohistochemical evaluation with caspase 3 antibody
Histological evaluation | one month
  Histological evaluation with Masson's trichrome dye

CONTACTS AND LOCATIONS:
Locations (1):
- Ibramed - Indústria Brasileira de Equipamentos Médicos, Amparo, São Paulo, Brazil